CLINICAL TRIAL: NCT05766735
Title: Treating Early Type 2 Diabetes by Reducing Postprandial Glucose Excursions: A Paradigm Shift in Lifestyle Modification
Acronym: GEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiara Fabris, PhD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chiara Fabris, PhD, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 220259; R01DK129687 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-03-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Routine Care (RC); Routine Care + Glycemic Excursion Minimization (RC+GEM); Continuous Glucose Monitor (CGM); Randomized Controlled Trial (RCT); Blood Glucose (BG); Newly Diagnosed Type 2 Diabetes; Type 2 diabetes (T2D); Primary Care Provider (PCP); Remote Study Visits
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to individualized routine care (RC) or to individualized RC in addition to post-nutrient glucose excursion minimization (RC+GEM). A Randomized Controlled Trial (RCT) design will be used to assign participants to treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (RC) (Active Comparator): Participants will be actively working with their primary care provider during the study and will attend appointments with their provider as needed. The study team will monitor their progress at the scheduled Assessment Visits. The participants should discuss any concerns they have, including side effects or cost, in order to adjust the medication regime with their primary care team. Their physician/clinician may recommend additional things, like weight loss, exercise programs and/or diabetes education programs.
  Interventions: Other: Routine Care (RC)
- Routine Care + Glucose Excursion Minimization (RC+GEM) (Experimental): Participants will actively work with their primary care provider and receive personalized routine care (RC). In addition, participants will receive GEM, an individualized, person-centered, empowerment program, not a behavior modification program. GEM provides individuals with personally relevant information to make choices that will help them achieve their diabetes goals. It focuses on techniques - eating low glycemic load foods, increasing moderate and vigorous exercise, and monitoring blood glucose (BG) to educate individuals about the impact of high glycemic load nutrients and vigorous exercise. The emphasis is on minimizing glucose excursions by any practical means, e.g., nutrient selection, timing and combinations of nutrient intake, time restricted eating, eating carbohydrates after protein and fat, post prandial physical activity, whatever is personally affirmed by BG feedback.
  Interventions: Behavioral: Routine Care + Glycemic Excursion Minimization (RC+GEM)

INTERVENTIONS:
Behavioral: Routine Care + Glycemic Excursion Minimization (RC+GEM) — In addition to receiving routine care, participants will receive GEM, a structured, self-directed, and personalized program that will allow participants with pre-diabetes to improve their metabolic status by illustrating the effects of their routine food and physical activity choices on their blood glucose levels and variability.
  Other Names: Glucose Everyday Matters
  Arms: Routine Care + Glucose Excursion Minimization (RC+GEM)
Other: Routine Care (RC) — RC participants will meet with their primary care provider to determine the best diabetes medication and proper dose. The participant will be allowed to change medications, or use a combination of medications, that is best suited for their care during the duration of the study. The study team will not influence these decisions.
  Arms: Routine Care (RC)

SUMMARY:
A Randomized Control Trial (RCT) with 1:1 randomization of adults newly diagnosed with type 2 diabetes (T2D) to Routine Care (RC) and RC + Glycemic Excursion Minimization (RC+GEM); a program that provides RC in addition to continuous glucose monitors (CGM) within a structured, self-directed, and personalized lifestyle program called GEM. Our hypothesis is that RC+GEM will: 1) reduce hemoglobin A1c as much or more, 2) require less diabetes medication, 3) cost less, and 4) have more secondary benefits, (e.g. greater reduction in cardiovascular risk, weight, diabetes distress, depression symptoms), compared to RC alone.

DETAILED DESCRIPTION:
The proposed study will compare individualized self-administered versions of RC+GEM to RC among patients recently diagnosed with type 2 diabetes. We hypothesize that, compared to RC alone, RC+GEM will be at least as effective at improving blood glucose control (A1c), and RC+GEM will do so with less reliance on diabetes medication and with greater secondary benefits such as lower risk of cardiovascular disease, more "good" cholesterol (HDL), greater weight loss, a greater sense of empowerment, and fewer diabetes-related expenses. It is further hypothesized that these benefits will be sustained over 13.5-months of follow-up with no structured maintenance program.

Remote study visits are permitted. Clinic visit and remote visits may include videoconferencing, phone, text messages and emails.

ELIGIBILITY:
Inclusion Criteria

1. Clinical diagnosis, based on investigator assessment, of type 2 diabetes within the past 24 months
2. Age ≥30.0 and ≤80 years
3. Hemoglobin A1c = ≥6.5-≤11% (medical record value <6 month-old is acceptable)
4. Access to smartphone throughout the study
5. Diabetes management visit with medical provider within 12 months of screening date
6. If on weight altering medications (e.g., GLP-1, GIP), on a stable dose for about four weeks

Exclusion Criteria:

1. Medications that impede weight loss within the last 3 months, per study physicians' discretion
2. Any psychotropic medication that could raise blood glucose, per study physicians' opinion
3. Conditions that preclude participating in the study (e.g., severe mental disease like manic depressive illness, severe depression, active substance abuse)
4. Conditions that preclude increasing physical activity (e.g., severe neuropathy, cardiovascular disease, COPD/emphysema, severe osteoarthritis, stroke)
5. Conditions that prevent doing the self-directed GEM program, such as inability to read English, mental health conditions that prevent engagement in treatment, such as active substance abuse, severe depression
6. Conditions that restrict diet such as severe gastroparesis, ulcers, or food allergies
7. Severe vision impairment that at PI discretion would preclude ability to read the GEM manual or see the information on the CGM or activity tracker
8. Currently undergoing treatment for cancer that in the opinion of the PI would preclude participation in the study
9. Renal impairment (for example eGFR < 45 mL/min/1.73 meters squared; CKD-3b)
10. Currently pregnant or contemplating pregnancy within the next 14 months
11. Currently breastfeeding
12. Any condition that, in the opinion of the principal investigator, could interfere with the safe and effective completion of the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c at 4.5-months of follow-up | 4.5 months
  Repeated measures models, using the baseline Hemoglobin A1c, as a covariate, will be used to compare groups with respect to Hemoglobin A1c levels at the 4.5-month assessment.
Change in Hemoglobin A1c at the 13.5-months of follow-up | 13.5 months
  Repeated measures models, using the baseline Hemoglobin A1c, as a covariate, will be used to compare groups with respect to Hemoglobin A1c levels at the 13.5-month assessment.
Change in Metformin at 4.5-months of follow-up | 4.5 months
  Repeated measures models, using baseline Metformin, as a covariate, will be used to compare groups with respect to Metformin at the 4.5-month assessment.
Change in Metformin at 13.5-months of follow-up | 13.5 months
  Repeated measures models, using baseline Metformin, as a covariate, will be used to compare groups with respect to Metformin at the 13.5-month assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Fabris, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology; Daniel J. Cox, PhD, AHPP, Principal Investigator — University of Virginia Center for Diabetes Technology; Tamara Oser, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Department of Family Medicine, Aurora, Colorado
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the publication of the manuscript.
Access Criteria: The Data Sharing Agreements will be formulated by the study team